CLINICAL TRIAL: NCT01206504
Title: Expanded Access to MGAWN1 in Subjects With: Suspected West Nile Neuroinvasive Disease; Suspected West Nile Virus Infection and a Compromised Immune System; or Substantial Accidental Exposure to West Nile Virus
Brief Title: Expanded Access to MGAWN1 in Subjects With Suspected West Nile Neuroinvasive Disease; Suspected West Nile Virus Infection; or Substantial Accidental Exposure
Status: No longer available | Type: Expanded Access
Sponsor: MacroGenics (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CP-MGAWN1-EA1
Record Dates: First submitted 2010-09-17; First posted 2010-09-22 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: West Nile Virus Infection
Keywords: West Nile virus; WNV; Encephalitis; Meningitis; Acute Flaccid Paralysis; Monoclonal Antibody; WNND; West Nile Neuroinvasive Disease; Accidental Exposure to West Nile Virus
MeSH Terms: conditions — West Nile Fever; Encephalitis; Meningitis; acute flaccid myelitis

INTERVENTIONS:
Biological: MGAWN1 — Humanized monoclonal to West Nile virus. Dose=30mg/kg

SUMMARY:
This study will test an experimental drug called MGAWN1 for the treatment of West Nile infections.

DETAILED DESCRIPTION:
The objective of this study is to provide expanded access to MGAWN1; the study is not intended for subjects who are eligible for and have access to non-expanded access protocols.

ELIGIBILITY:
Inclusion Criteria:

1. For West Nile Neuroinvasive Disease subjects: Have neurological signs and/or symptoms of West Nile meningitis, encephalitis, and/or acute flaccid paralysis
2. For immunocompromised subjects with suspected West Nile virus infection:

   * Receiving immunosuppressive treatment for any disease, such as autoimmune diseases, or transplant recipients; or
   * Have received organs or tissues or cells from donors likely infected with West Nile virus (as shown by serology or PCR/NAT from the donor, organs, or tissues) or
   * Have acquired immunodeficiency (other than from immunosuppressive treatment or from receiving infected transplants) or congenital immunodeficiency
3. For subjects with substantial exposure to West Nile virus: Exposure by any route, including percutaneous, inhalation, or mucosal exposure (such as might occur in a laboratory accident)
4. Develop signs and/or symptoms within 14 days before study enrollment

Min Age: 8 Years | Sex: All
Age Groups: Child, Adult, Older Adult